CLINICAL TRIAL: NCT01976169
Title: Phase 1B Study of PD-0332991 in Combination With T-DM1 in the Treatment of Patients With Advanced HER2 (Human Epidermal Growth Factor Receptor 2)-Positive Breast Cancer
Brief Title: Phase 1b Study of PD-0332991 in Combination With T-DM1(Trastuzumab-DM1)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Pfizer (Industry); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 042013-042
Record Dates: First submitted 2013-10-29; First posted 2013-11-05 (Estimated); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Advanced Breast Cancer
Keywords: Breast Cancer; Advanced Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; Ado-Trastuzumab Emtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PD-0332991 and T-DM1 (Experimental): The subjects will be administered T-DM1 by intravenous infusion at 3.6 mg/kg for 90 minutes on day 1 of each 21 day cycle. Infusion timing may vary from 30-90 minutes depending on how well the subject tolerates the treatment.
  A standard 3+3 trial design will be used for PD-0332991 dose escalation cohorts.The dosing of PD-0332991 will be divided into 3 cohorts, the subjects will receive PD-0332991 on days 5-18 of each 21 day cycle.
  Cohort 1 : PD-0332991 - 100 mg daily (oral) Cohort 2 : PD-0332991 - 150 mg daily (oral) Cohort 3 : PD-0332991 - 200 mg daily (oral)
  Interventions: Drug: PD-0332991 and T-DM1

INTERVENTIONS:
Drug: PD-0332991 and T-DM1 — The subjects will be administered T-DM1 by intravenous infusion at 3.6 mg/kg for 90 minutes on day 1 of each 21 day cycle. Infusion timing may vary from 30-90 minutes depending on how well the subject tolerates the treatment.
  A standard 3+3 trial design will be used for PD-0332991 dose escalation cohorts.The dosing of PD-0332991 will be divided into 3 cohorts, the subjects will receive PD-0332991 on days 5-18 of each 21 day cycle.
  Cohort 1 : PD-0332991 - 100 mg daily (oral) Cohort 2 : PD-0332991 - 150 mg daily (oral) Cohort 3 : PD-0332991 - 200 mg daily (oral)
  Other Names: KADCYLA=T-DM1; Palbociclib=PD-0332991

SUMMARY:
Standard of care:

Treatment with Trastuzumab

Experimental:

21-Day Cycle of Combination therapy with T-DM1 intravenously on Day 1 and oral PD-0332991 on Days 5-18

Study Design and Methodology:

This is a phase 1B inter-patient dose escalation study of PD-0332991 in combination with T-DM1 in patients with recurrent or metastatic HER2-positive breast cancer after prior trastuzumab or other HER2-directed therapies.

The subjects will be administered T-DM1 by intravenous infusion at 3.6 mg/kg for 90 minutes on day 1 of each 21 day cycle. Infusion timing may vary from 30-90 minutes depending on how well the subject tolerates the treatment.

A standard 3+3 trial design will be used for PD-0332991 dose escalation cohorts.The dosing of PD-0332991 will be divided into 3 cohorts, the subjects will receive PD-0332991 on days 5-18 of each 21 day cycle.

Cohort 1 : PD-0332991 - 100 mg daily (oral) Cohort 2 : PD-0332991 - 150 mg daily (oral) Cohort 3 : PD-0332991 - 200 mg daily (oral)

The 3+3 design entails that if one patient out of the first three patients has a DLT, up to three additional patients will be entered at that dose level

Treatment cycles will continue until disease progression or withdrawal from study.

DETAILED DESCRIPTION:
This is a phase 1B inter-patient dose escalation study of PD-0332991 in combination with T--DM1 in patients with recurrent or metastatic HER2-positive breast cancer after prior trastuzumab or other HER2-directed therapies. A standard 3+3 trial design will be used for PD-0332991 dose escalation cohorts. The 3+3 design entails that if one patient out of the first three patients has a dose-limiting toxicity (DLT), three additional patients will be entered at that dose level. The PD-0332991 dose levels will start at 100 mg po daily; the second cohort will receive 150mg po daily; the third cohort 200mg po daily. Patients receive PD-0332991 on days 5-18 of each 21 day cycle. T-DM1 will be given intravenously at 3.6 mg/kg on day 1 of each 21 day cycle.

Toxicity will be assessed using the Common Terminology Criteria of Adverse Events (CTCAE) version 4.0 grading scale. Dose- limiting toxicity-DLT is defined as any drug-related grade 3 non-hematologic toxicity or grade 4 hematologic toxicity lasting >28 days after the last day of therapy. If two patients experience drug-related DLT, the maximal tolerated dose (MTD) for the combination in HER2-positive breast cancer patients has been exceeded, enrollment to that dose will stop, and the next lower dose will be designated the MTD. An additional 15 patients will be treated at the MTD or the maximal 200mg po daily PD-0332991 dose in combination with T-DM1 to confirm safety. Treatment cycles will continue until disease progression or withdrawal from study.

Study End-points:

1. To evaluate and assess Dose Limiting Toxicities (DLT).
2. To determine the toxicity profile.
3. To determine the clinical response rate.
4. To determine the duration of response.
5. To evaluate baseline HER2 positivity biomarkers by analyzing pretreatment tumor Ki67, phospho-RB, cleaved caspase 3, phospho-histone H3, cycline E, MCM7, HER2, p27Kip1.
6. To evaluate post-treatment Ki67, phospho-RB, cleaved caspase 3, phospho-histone H3, cyclin E, MCM7, HER2, p27Kip1, Rb, p16ink4c, CDK4, CDK6 in order to establish biomarker response to treatment.
7. To evaluate pharmacokinetic (PK) parameters for PD-0332991 and T-DM1 including Cmax, AUC, t1/2

ELIGIBILITY:
Inclusion Criteria:

* 1.All subjects must be informed about the study and have signed a current IRB (Institutional Review Board) approved informed consent.

  2. All subjects must have recurrent or metastatic HER2-positive breast cancer. diagnosed by biopsy.

  3. All subjects must have previously received trastuzumab or other HER2 targeted therapies.

  4.Tumor must be HER2-positive and RB-proficient. RB (Retinoblastoma protein)-proficiency is determined by tumor biopsy demonstrating RB normal and p16in4a low by immunohistochemistry. RB proficiency means that there is an intact RB pathway indicative of responsiveness to PD-0332991. RB staining is scored on an absent (no nuclear staining), weak (nuclear staining less than observed in endothelial cells and stromal cells surrounding the tumor), positive (nuclear staining at or above surrounding tissue) (0, 0.5, 1 respectively). P16ink4a is a routine clinical stain that is scored using absent, weak, positive, strong (0,1,2,3 respectively). Tumors will be scored using [p16]/[RB], where a score of less than 3 is required for inclusion. RB loss is expected to occur in less than 15% of cases.

  5. Subjects must have a performance status of ≤ 2 on the ECOG (Eastern Cooperative Oncology Group)Performance scale.

  6. Subjects must have bilirubin <1.5 mg/dl, transaminases <2.5x upper limit of normal, albumin >3gm/dl, creatinine <1.3mg/dl, adequate cardiac reserve (EF>50%), ANC (Absolute neutrophil count) >1,000/mcL (microliter), and Platelets >100,000/mcL.

  7. Must be willing to be treated at the University of Texas Southwestern Hospital, University of Pennsylvania and affiliated clinics.

  8. Subjects must be willing to use an approved form of birth control while on this study and for 90 days after completion.

  9. Age > 18 years. 10. Subject must be able to swallow capsules and have no surgical or anatomic condition that will preclude the subject from swallowing and absorbing oral medications on an ongoing basis.

Exclusion Criteria:

* 1. Chemotherapy, radiotherapy or hormonal therapy within 3 weeks ( 6 weeks for nitrosoureas, mitomycin C or bevacizumab), or who have not recovered from the adverse events to < grade 2 due to previous agents administered more than 4 weeks prior to Study Day 1.

  2. Subjects less than 4 weeks post major surgery. 3. Known active CNS metastases or carcinomatous meningitis. Subjects with CNS (Central Nervous System) metastases including brain metastases who have completed a course of radiotherapy are eligible for the study provided they are clinically stable. However, oral corticosteroids for control of CNS symptoms are not allowed.

  4. Known documented or suspected hypersensitivity to the components of the study drug(s) or analogs.

  5. Uncontrolled systemic illness, including but not limited to ongoing or active infection.

  6. Symptomatic congestive heart failure, unstable angina pectoris, stroke or myocardial infarction within 3 months.

  7. Baseline neuropathy >grade 1. 8. Known positive for human immunodeficiency virus (HIV). Baseline HIV screening is not required.

  9. Pregnant or breast-feeding subjects. 10. Subjects who are unable or unwilling to abide by the study protocol or to cooperate fully with the investigator or designee.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-01-24 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2021-05-19 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 42 days at the end of Cycle 2
  A standard 3+3 trial design will be used for PD-0332991 dose escalation cohorts.The dosing of PD-0332991 will be divided into 3 cohorts, the subjects will receive PD-0332991 on days 5-18 of each 21 day cycle.
  Cohort 1 : PD-0332991 - 100 mg daily (oral) Cohort 2 : PD-0332991 - 150 mg daily (oral) Cohort 3 : PD-0332991 - 200 mg daily (oral)
Dose Limiting Toxicities (DLT) | 42 days at the end of Cycle 2
  The 3+3 design entails that if one patient out of the first three patients has a DLT, up to three additional patients will be entered at that dose level

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Haley, MD, Principal Investigator — Internal Medicine Hematology Oncology
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No